CLINICAL TRIAL: NCT07308925
Title: Effectiveness of Using Real-time Continuous Glucose Monitoring Compared With Intermittent Continuous Glucose Monitoring in People With Type 2 Diabetes Treated With Insulin.
Brief Title: Real-time Continuous Glucose Monitoring Compared With Intermittent Continuous Glucose Monitoring in People With Type 2 Diabetes Treated With Insulin.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario San Ignacio (Other)
Collaborators: Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FM-CIE-1013-24
Record Dates: First submitted 2025-09-20; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Continuous Glucose Monitoring; Time in Range
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: open-label randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- isCGM (No Intervention): Usual Care + isCGM Group: Patients in this group will have the FreeStyle Libre 2 continuous interstitial glucose monitoring sensor (Abbott Diabetes Care Inc., Alameda, CA, USA) inserted. High glucose alarms (>250 mg/dL) and low glucose alerts (<70 mg/dL) will be programmed. They will also be instructed to perform at least eight scans daily to avoid data loss. All participants were instructed to replace their sensors according to the manufacturer's recommendations: every 15 days for isCGM.
- RT-CGM (Experimental): • Usual care + TR-CGM group: Patients in this group will undergo insertion of a continuous interstitial glucose monitoring (CGM) sensor using the FreeStyle Libre 2 Plus device and LibreLink app® (Abbott Diabetes Care, Inc., Alameda, CA, USA). The sensor will be programmed with high glucose alarms (>250 mg/dL) and low glucose alerts (<70 mg/dL). All participants will be instructed to replace their sensor according to the manufacturer's recommendations: every 15 days for TR-CGM.
  Interventions: Device: real time Continuous Glucose Monitoring

INTERVENTIONS:
Device: real time Continuous Glucose Monitoring — • Usual care + TR-CGM group: Patients in this group will undergo insertion of a continuous interstitial glucose monitoring (CGM) sensor using the FreeStyle Libre 2 Plus device and LibreLink app® (Abbott Diabetes Care, Inc., Alameda, CA, USA). The sensor will be programmed with high glucose alarms (>250 mg/dL) and low glucose alerts (<70 mg/dL). All participants will be instructed to replace their sensor according to the manufacturer's recommendations: every 15 days for TR-CGM.
  Other Names: RT-CGM
  Arms: RT-CGM

SUMMARY:
The objective is to compare the efficacy of TR-CGM versus isCGM in patients diagnosed with T2D who are treated with insulin and use CGM, as defined by time in range between 70 and 180 mg/dL.

An open-label clinical trial will be conducted. Patients with T2D who use intermittent glucose monitoring and insulin with poor metabolic control will be included. They will be randomized to continue with isCGM or RT-CGM.

The primary outcome: %TIR 70-180 mg/dL.

DETAILED DESCRIPTION:
All patients diagnosed with type 2 diabetes (T2D) who meet the inclusion criteria will be identified (see inclusion and exclusion criteria). They will then be invited to participate in the study and asked to sign an informed consent form. Demographic data, baseline clinical characteristics, and clinical tests related to metabolic control will be collected.

Visit 0 (V0): Informed consent signature and basal CGM system installation will be verified.

Visit 1 (V1): CGM data will be downloaded. All enrolled patients will receive the same instructions for device use and management of high and low glucose levels, according to standard clinical procedures. Then, randomization will be performed by someone who is blinded to the clinical characteristics of each patient and is not part of the research group. The allocation given by this mechanism cannot be changed by the treating physicians.

* Usual care + TR-CGM group: Patients in this group will receive a continuous interstitial glucose monitoring (CIGM) sensor via the FreeStyle Libre 2 Plus device and LibreLink app® (Abbott Diabetes Care, Inc., Alameda, CA). High alarms greater than 250 mg/dL and low glucose alerts less than 70 mg/dL will be programmed. All participants will be instructed to change their sensor according to the manufacturer's recommendations: every 15 days for the TR-CGM group.
* Usual care + CIGM group: Patients in this group will receive a CIGM sensor using the FreeStyle Libre 2 device (Abbott Diabetes Care Inc., Alameda, CA, USA). High alarms >250 mg/dL and low glucose alerts <70 mg/dL will be programmed. Additionally, they will be instructed to perform at least eight scans daily to avoid data loss. All participants were instructed to change their sensors according to the manufacturer's recommendations: every 15 days for isCGM.

Standard Care (Applies to Both Groups):

All patients should be assessed by the diabetes clinic's nutrition service, which will provide basic dietary and physical activity recommendations.

All patients will be instructed in basal and/or prandial insulin titration, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 35 years.
* HbA1c >7.0%
* Treatment with one or more insulin injections.
* Stable medication regimen for the 3 months prior to study entry.
* Insulin treatment for ≥3 months with a stable dose prior to entry, with fasting blood glucose between 70 and 130 mg/dL.
* Availability of an NFC-enabled smartphone.

Exclusion Criteria:

* Pregnancy or planning to become pregnant during the study period.
* History of bariatric surgery within the year prior to study entry or plans to undergo bariatric surgery during the study.
* Having a condition that would likely require an MRI during the study period.
* Use of medications containing high doses of ascorbic acid (>2000 mg/day), as it may falsely increase sensor readings.
* Concomitant illness or condition that may compromise patient safety, including, but not limited to, serious mental illness, a diagnosed or suspected eating disorder, or any long-term medical/unmanageable disorder.
* GFR less than 30 ml/min.
* Psychiatric condition that interferes with study-related tasks.
* Known (or suspected) significant allergy to medical-grade adhesives.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Time in Range | 12 weeks
  To compare the efficacy defined as time in range between 70 - 180 mg/dl of the TR-CGM compared to isCGM in patients diagnosed with T2DM treated with insulin who use CGM as part of usual clinical practice in follow-up at the endocrinology unit of the San Ignacio University Hospital.

SECONDARY OUTCOMES:
Proportion of patients with a ≥5% increase in TIR | 12 weeks
  Compare the proportion of patients with a ≥5% increase in TIR 70-180 mg/dl compared to the initial value.
TAR | 12 weeks
  To compare percentage of time in hyperglycemia range >180 and >250 mg/dl
TBR <70 mg/dl | 12 weeks
  To compare the proportion of patients with a %TBR <70 mg/dL to less than 4%
TBR <54 mg/dl | 12 weeks
  To compare the proportion of patients with a %TBR <54 mg/dL to less than 1%
Severe hypoglycemia | 12 weeks
  To compare the incidence of severe hypoglycemia, hospitalizations, and emergency department visits.
Satisfaction with the device | 12 weeks
  To compare satisfaction with the device using the "Questionnaire on experience with glucose monitoring (C-EMC)" at the end of the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Diana C Henao-Carrillo, Endocrinologyst, Principal Investigator — Hospital Universitario San Ignacio
Locations (1):
- Hospital Universitario San Ignacio, Bogotá, Colombia